CLINICAL TRIAL: NCT06484777
Title: An Open-label, Multi-center Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of SHR-9539 Injection in Patients With Multiple Myeloma
Brief Title: A Clinical Study of SHR-9539 in Patients With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-9539-101
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-9539 for injection (Experimental)
  Interventions: Drug: SHR-9539 for injection

INTERVENTIONS:
Drug: SHR-9539 for injection — SHR-9539 for dose escalation/dose extension

SUMMARY:
This study is a multicenter, open-label, dose-escalation/dose-expansion clinical Phase I trial designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy profile of SHR-9539 Injection in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on day of signing the Informed Consent Form;
2. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale；
3. Documented initial diagnosis of multiple myeloma according to IMWG diagnostic criteria ；
4. Have a life expectancy of at least 3 months；
5. Male and female subjects with fertility must agree to use efficient contraceptive measures with their partners within 3 months after the last administration of the test drug from the time of signing the informed consent form, and have no fertility plan and avoid donating sperm / eggs. The pregnancy test during the screening period must be negative.

Exclusion Criteria:

1. Central nervous system (CNS) involvement of MM；
2. Diagnosis of amyloidosis, plasma cell leukemia, Wahl's macroglobulinemia, or POEMS syndrome;
3. Prior Grade 3 or higher CRS (Per ASTCT standards) related to any T cell redirection (eg, CD-3 redirection technology or CAR-T cell therapy).
4. Have other factors that may force the termination of the study, e.g., non-compliance with the protocol, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory abnormalities, associated family or social factors, which would affect the safety of the subjects or the collection of data and samples, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
RP2D of SHR-9539 injection | Approximately 24 months
  Determination of the recommended phase 2 dose (RP2D) of SHR-9539 injection in patient with multiple myeloma.

SECONDARY OUTCOMES:
Incidence and severity of AE | Up to follow-up period, approximately 24 months
  Assessing the incidence of adverse events (AEs) mainly using the Common Terminology Criteria for Adverse Events (CTCAE Version 5), and CRS and ICANS were graded according to ASTCT standards.
Cmax | Up to follow-up period, approximately 24 months
  Maximum serum concentration
Tmax | Up to follow-up period, approximately 24 months
  Time to reach maximum plasma concentration.
Overall Response Rate (ORR) | Up to follow-up period, approximately 24 months
  ORR assessed by the IMWG response criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided